CLINICAL TRIAL: NCT02179073
Title: Effects of Bladder Management on Health-related Quality of Life in Patients With Neurogenic Bladder
Brief Title: Health-related Quality of Life of Patients With Neurogenic Bladder
Status: Completed | Type: Observational
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Other Study IDs: 2007-02
Record Dates: First submitted 2014-06-26; First posted 2014-07-01 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Neurogenic Bladder Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- neurogenic bladder dysfunction

SUMMARY:
Bladder management has a major impact on the quality of life in patients with neurogenic bladder dysfunction. This a prospective investigation of the effects of the method for bladder evacuation on the health-related quality of life in patients with neurogenic bladder dysfunction. The changes in health-related quality of life over time (longitudinal investigation) and the differences between the different methods for bladder evacuation will be investigated. Patients will be given a standardized and validated questionnaire annually for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with neurogenic bladder dysfunction

Exclusion Criteria:

* Insufficient dexterity to fill in the questionnaire
* Insufficient proficiency in the German or French language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: individuals with neurogenic bladder dysfunction
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2007-12; Primary Completion 2019-10-31 (Actual); Study Completion 2019-11-14 (Actual)

PRIMARY OUTCOMES:
quality of life | up to year 10
  Qualiveen questionnaire

SECONDARY OUTCOMES:
bladder evacuation method | year 1, 2, 3, 4, 5, 6, 7, 8, 9, 10
  method for bladder evacuation (i.e. intermittent catheterization, condom urinal, reflex micturition, transurethral catheter, suprapubic catheter, sacral bladder stimulator, neuromodulation)
urinary tract infections | year 1, 2, 3, 4, 5, 6, 7, 8, 9, 10
  number of annual symptomatic urinary tract infections
patient characteristics | time 0
  gender, age, type of neurogenic bladder dysfunction, duration of neurogenic bladder dysfunction

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland